CLINICAL TRIAL: NCT02971553
Title: A Randomised Controlled Trial on Positive End-expiratory Pressure (PEEP) During Resuscitation of Non-breathing Neonates
Brief Title: PEEP Resuscitation Trial
Acronym: PEEPrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haydom Lutheran Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Upright PEEP
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Newborn Resuscitation
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upright Resuscitator with PEEP (Experimental): Ventilation with the Upright Resuscitator with PEEP
  Interventions: Device: Upright Resuscitator with PEEP
- Upright Resuscitator (Active Comparator): Ventilation with the Upright Resuscitator (without PEEP)
  Interventions: Device: Upright Resuscitator

INTERVENTIONS:
Device: Upright Resuscitator with PEEP
  Arms: Upright Resuscitator with PEEP
Device: Upright Resuscitator
  Arms: Upright Resuscitator

SUMMARY:
Each year, almost 3 million newborn babies die within their first month of life, often as a consequence of labour complications. Approximately 5% of newborns will not start breathing at birth and need immediate help. The optimal ventilation strategy with liquid-filled lungs has not been determined. Animal studies suggest that assisted ventilation with positive end expiratory pressure (PEEP) improves the aeration of liquid-filled lungs leading to more rapid recovery. However, no large human clinical studies have investigated the clinical responses to assisted ventilation with PEEP in asphyxiated newborns.

DETAILED DESCRIPTION:
Laerdal Global Health has developed a PEEP valve which has been tested and shown to provide reliable end-expiratory pressures in a manikin model, even with a high mask leak. Whether this PEEP valve provides reliable PEEP in vivo and whether this translates to clinical beneficial outcomes remains to be proven.

The aim is to study whether lung aeration can be improved by adding a device for positive end expiratory pressure (PEEP) to better distend the airways in neonates more than 28 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who need assisted bag/mask ventilation after birth due to failure to initiate breathing the first 60 seconds after birth.

Exclusion Criteria:

* Babies with major deformities not deemed to be viable.
* Missing parental consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Delta heart rate (beats/minute) during each ventilation sequence | 10 minutes

SECONDARY OUTCOMES:
Neonatal outcome dead versus alive | Up to 24 hours
Time to cessation of ventilation | Up to 1 hour
Time to heart rate above 140 beats/minute | Up to 1 hour
Mean ariway pressures given | Up to 1 hour
Time to detection of exhaled CO2 above 1% and 4% | Up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Kidanto, MD, PhD, Principal Investigator — Muhimibili National Hospital
Locations (1):
- Haydom Lutheran Hospital, Research Institute, Haydom, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holte K, Ersdal H, Eilevstjonn J, Gomo O, Klingenberg C, Thallinger M, Linde J, Stigum H, Yeconia A, Kidanto H, Stordal K. Positive End-Expiratory Pressure in Newborn Resuscitation Around Term: A Randomized Controlled Trial. Pediatrics. 2020 Oct;146(4):e20200494. doi: 10.1542/peds.2020-0494. Epub 2020 Sep 11. PMID 32917847